CLINICAL TRIAL: NCT04412330
Title: Optimizing Outcomes With Physical Therapy Treatment for IndividuALs Surviving an ICU Admission for Covid-19 (OPTImAL) - a Single Center Prospective Study
Brief Title: Optimizing Outcomes With Physical Therapy Treatment for IndividuALs Surviving an ICU Admission for Covid-19
Acronym: OPTIMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: Ashley Montgomery-Yates (Unknown)
Responsible Party: Principal Investigator, Kirby Mayer, Assistant Professor, University of Kentucky
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59097
Record Dates: First submitted 2020-05-12; First posted 2020-06-02 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Covid-19; Critical Illness; Post Intensive Care Unit Syndrome; Muscle Weakness
MeSH Terms: conditions — COVID-19; Critical Illness; Muscle Weakness | interventions — Physical Therapy Modalities

STUDY DESIGN:
Masking Description: Prospective study with one-treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICU followup + physical therapy (Experimental): Patients surviving ICU admission for Covid-19 will receive ICU follow-up care in an ICU Recovery Clinic plus 8 weeks of physical therapy interventions. ICU Recovery Clinic is standard of care for patients surviving medical ICU admission at University of Kentucky with potential to attend in person or complete through telemedicine up to 5 appointments in the first year after hospital discharge. Physical therapy interventions completed at an outpatient pulmonary rehabilitation center or through telemedicine is not currently standard of care for patients in the short-term recovery phase (1-6 months after hospital discharge) after critical illness.
  Interventions: Other: ICU Recovery + Physical Therapy

INTERVENTIONS:
Other: ICU Recovery + Physical Therapy — Physical therapy interventions will be supervised by a physical therapist (>20 years of experience in ICU and pulmonary rehabilitation). Potential interventions include endurance/aerobic training (treadmill training, upper and lower extremity ergometer, and recumbent step machine), upper and lower extremity resistance strength training, balance training, functional movement training, and education. If the interventions are providing in the home environment the exercises will be completed through Zoom, video communications app. Home-based interventions will include seated and standing exercise including resistance exercises (such as lifting small weights) and endurance (e.g. marching or stepping in place, repetitive sit-to-stand training). Physical therapist will provide verbal instructions for motivation and adherence to exercise interventions.

SUMMARY:
Introduction: Survivors of acute respiratory failure develop persistent muscle weakness and deficits in cardiopulmonary endurance combining to limit physical functioning. Early data from the Covid-19 pandemic suggest a high incidence of critically ill patients admitted to intensive care units (ICU) will require mechanical ventilation for acute respiratory failure. Covid-19 patients surviving an admission to the ICU are expected to suffer from physical and cognitive impairments that will limit quality of life and return to pre-hospital level of functioning. In this present study, the investigators will evaluate the safety and feasibility of providing a novel clinical pathway combining ICU after-care at an ICU Recovery clinic with physical therapy interventions.

Methods and Analysis: In this single-center, prospective (pre, post cohort) trial in patients surviving ICU admission for Covid-19. The investigators hypothesize that this novel combination is a) safe and feasible to provide for patients surviving Covid-19; b) improve physical function and exercise capacity measured by performance on 6-minute walk test and Short Performance Physical battery; and c) reduce incidence of anxiety, depression and post-traumatic stress assessed with Hospital Anxiety and Depression Scale and the Impact of Events Scale-revised. Safety will be assessed by pooled adverse events and reason for early termination of interventions. Feasibility will be assessed by rate of adherence and attrition. Repeated measures ANOVA will be utilized to assess change in outcomes from at first ICU Recovery Clinic follow-up (2-weeks) and 3- and 6-months post hospital discharge.

Ethics and Dissemination: The trial has received ethics approval at the University of Kentucky and enrollment has begun. The results of this trial will support the feasibility of providing ICU follow-up and physical therapy interventions for patients surviving critical illness for Covid-19 and may begin to support effectiveness of such interventions. Investigators plan to disseminate trial results in peer-reviewed journals, as well as presentation at physical therapy and critical care national and international conferences.

DETAILED DESCRIPTION:
ICU Recovery Clinic is standard of care for patients surviving a critical illness in the Medical ICU at the University of Kentucky. The ICU Recovery Clinic includes a transdisciplinary team with input from five disciplines that provide coordinated outpatient care with a focus on medical issues, medication management, nutrition, sleep disruption, and any issues related to post-intensive care syndrome such as anxiety, depression, PTSD, cognitive dysfunction and physical impairments.

Individualized physical therapy treatment: After the initial ICU recovery clinic appointment patients will begin their 8-week physical therapy program which will be delivered 1-2 times per week in a supervised 1:1 session and supplemented with 3 days of unsupervised home exercises and walking program on days not participating in physical therapy sessions. Supervised sessions will be run by a physical therapist (>20 years of experience in ICU and pulmonary rehabilitation) either face to face in outpatient setting or through telemedicine using video consultation platforms for patients unable to attend appointments due to transmission risk, transportation issues, or geographically living >45 miles from clinic. Prior to commencing the first treatment session patients will complete baseline testing to inform the starting parameters (frequency, intensity, repetitions) based on performance in physical tests such as 6MWT and muscle strength testing. The patient will receive an individualized and tailored physical therapy treatment, which will be targeted towards increasing their aerobic fitness, muscle strength and functional ability.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age) surviving an ICU admission with laboratory confirmed Covid-19.

Exclusion Criteria:

* pre-existing neurological or orthopedic injury, disease, or condition that would prevent participation in exercise interventions.
* patient not ambulatory prior to hospitalization
* patient not expected to survivor 90 days after hospitalization
* pregnant
* prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Adverse events (safety) | through study completion, an average of 3-months
  Incidence of adverse events, quantified by pain or discomfort that causes termination of interventions; a fall (with or without injury) during interventions or directly related to interventions such as fall due to fatigue; and physiologic event/abnormality that warrants termination of interventions or medical follow-up including bradycardia, tachycardia, and emergent hypertension

SECONDARY OUTCOMES:
Feasibility (success of consent process, adherence, and attrition) | through study completion, an average of 3-months
  Feasibility will be assessed by the consent rate (number of patients agreed to participate/number of patients approached for consent) and adherence attendance measured by the percentage of sessions patient participated divided total number of scheduled appointments. Adherence will also be prospectively assessed by total duration of exercise, dosage and intensity of exercises as described above. Attrition will be quantified by number of patients lost to follow-up.
Six minute walk test | Assessed at baseline, and repeated 3- and 6-months post hospital discharge
  Distance walked on six-minute walk test performed in line with the ATS/ERS Guidelines as measure of exercise capacity
Short Performance Physical Battery | Assessed at baseline, and repeated 3- and 6-months post hospital discharge
  Short Performance Physical Battery (SPPB) is a performance-based physical function test with components of balance, repetitive five times sit-to-stand for time, and 4-meter habitual gait speed. Higher scores on SPPB indicate better physical function.
Quality of life (EQ-5DL) | Assessed at baseline, and repeated 3- and 6-months post hospital discharge
  Health-related quality of life (HRQoL) will be measured by self-report questionnaire, the Five Dimension Euro-Quality of Life (EQ-5D) that includes a visual analog scale with rating for overall HRQoL (0-100)
Cognitive function | Assessed at baseline, and repeated 3- and 6-months post hospital discharge
  Cognitive function will be assessed by the Montreal Cognitive Assessment (MOCA) with <23/30 distinguishing mild cognitive impairment. If the patient participating in telemedicine through Zoom then the MOCA-Blind version will be completed.
Anxiety and Depression | Assessed at baseline, and repeated 3- and 6-months post hospital discharge
  Anxiety and depression will be assessed with the Hospital Anxiety and Depression Scale (HADS), a fourteen-item scale with subset scores of >8/21 indicating anxiety or depression
PTSD and distress | Assessed at baseline, and repeated 3- and 6-months post hospital discharge
  Distress and Post-traumatic stress disorder (PTSD) will be assessed through the Impact of Events Scale-Revised (IES-R), a 22-item self-report measure, with scores >35/88 recommending provisional diagnosis of PTSD
Return to work | Assessed at baseline, and repeated 3- and 6-months post hospital discharge
  For patients previously employed, the return to work will be assessed using the self-report survey instrument designed for ICU follow-up
Secondary complication | Assessed 3 and 6-months post hospital discharge
  Readmission rate and morality with be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Kirby P Mayer, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No